CLINICAL TRIAL: NCT03500835
Title: An Addiction Model Based Mobile Health Weight Loss Intervention With Coaching in Adolescents With Overweight and Obesity: Multi-Site Randomized Controlled Trial
Brief Title: An Addiction-Based Mobile Health Weight Loss Intervention With Coaching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: Cedars-Sinai Medical Center (Other); University of California, Los Angeles (Other); Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Principal Investigator, Alaina P. Vidmar, MD, Assistant Professor Department of Pediatric Endocrinology, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CHLA-18-00134
Record Dates: First submitted 2018-04-10; First posted 2018-04-18 (Actual); Results first posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-10

CONDITIONS: Pediatric Obesity; Mobile Technology; Addiction
MeSH Terms: conditions — Pediatric Obesity; Behavior, Addictive | interventions — Amyloid

STUDY DESIGN:
Intervention Model Description: The proposed multi-site randomized control trial (RCT) will test the effectiveness of an addiction-based weight loss intervention, embodied as a smartphone app with telephone coaching compared 1) an addiction-based weight loss intervention alone and 2) an in-clinic weight management intervention based on a traffic-light based approach in a larger sample of economically, racially and ethnically diverse adolescents (ages 14-18).
Who Masked: Outcomes Assessor
Masking Description: Blocked randomization will be utilized, to ensure the groups are balanced in terms of number of subjects and the distribution of potential confounding variables. Blocked randomization will be used to ensure the number of eligible subjects assigned to each group is equally distributed. Block size will be blinded from the primary investigator performing the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- App Plus Coaching (AC) (Experimental): 6 month addiction model based weight loss intervention in the form of an iPhone app coupled with personalized coaching.
  Interventions: Behavioral: App; Behavioral: Coaching
- App Alone (AA) (Experimental): 6 month addiction model based weight loss intervention in the form of an iPhone app.
  Interventions: Behavioral: App
- Clinic (Experimental): In-Clinic Multi-disciplinary monthly weight management program. Curriculum adapted from the KidsNFitness Program and administered by an MD, RD, Psychologist and Health Educator over 90 minute sessions
  Interventions: Behavioral: Clinic: Modified KidsNFitness

INTERVENTIONS:
Behavioral: App — 1. 6 month app intervention: Problem Food Withdrawal, Snacking Elimination and Food Amount Reduction
  2. Daily Weigh In
  3. App based reminders
  4. Follow Up: Face-to-face clinic visits at 3,6,12 and 18 months.
  Arms: App Alone (AA); App Plus Coaching (AC)
Behavioral: Coaching — 1. 6 month addiction based intervention: Problem Food Withdrawal, Snacking Elimination and Food Amount Reduction.
  2. Daily Weighing
  3. Daily Text messages from Coach
  4. Weekly 15 minute phone meetings with Coach
  5. Follow Up: Face-to-face clinic visits at 3,6,12 and 18 months post consent
  Arms: App Plus Coaching (AC)
Behavioral: Clinic: Modified KidsNFitness — 1. 6 month in-clinic, evidence-based, multi-disciplinary intervention
  2. 90 minute sessions, in clinic that occur every month for 6 months
  3. Follow Up: Face-to-face clinic visits Monthly x 6 months followed by face-to-face visit at12 and 18 months.
  Arms: Clinic

SUMMARY:
The proposed multi-site randomized control trial (RCT) will test the effectiveness of an addiction-based weight loss intervention, embodied first as a smartphone app with telephone coaching and second as an identical approach phone-coaching alone intervention compared to age matched controls participating in an in-clinic weight management interventions in a larger sample of economically, racially and ethnically diverse adolescents (ages 14-18). One hundred and eighty adolescents will be recruited from pediatric interdisciplinary weight management clinics operating out of five different hospital systems in Southern California and through targeted mailing to 40 ethnically, racially and economically diverse neighborhoods in Los Angeles County. The adolescents will be randomized 1:1 via stratified block randomization to either receive 1) interactive addiction model based mobile health (mHealth) weight-loss intervention with personalized phone-coaching (AppCoach), 2) interactive addiction model based mHealth weight-loss intervention alone (App) or 3) Multidisciplinary in-clinic weight management program (Clinic). Assessment of the intervention's effect on zBMI and percent over the 95th percentile (%BMIp95), fasting metabolic parameters, addictive eating habits, executive function, and motivation for change will be obtained at enrollment, 3, 6, 12 and 18 months (1 year post intervention follow up).

DETAILED DESCRIPTION:
Aim 1 (Primary Outcomes): To test the effectiveness of an addiction-based weight loss intervention, embodied first as a smartphone app with telephone coaching (AppCoach) compared to (1) addiction model based weight-loss app alone (App) and (2) multi-disciplinary in-clinic weight loss intervention (Clinic) on weight outcomes of overweight and obese adolescents at 3, 6, 12 and 18 months post enrollment.

Hypothesis 1a: Participants who complete the six month AppCoach will have a greater decrease in their zBMI and %BMIp95 compared to baseline at completion of the 6 months intervention, than those receiving App or Clinic.

Hypothesis 1b: Participants who completed the six month AppCoach will have greater decrease in their zBMI and %BMIp95 compared to baseline at 6 and 12 months post intervention completion compared to App and Clinic.

Aim 2 (Secondary Outcomes): To compare the effects of AppCoach on addictive eating behaviors, motivation and self-regulatory behaviors at completion of the intervention and 6 and 12 months post intervention.

Hypothesis 2: Compared to App or Clinic, AppCoach will result in lower YFAS-c scores, higher motivation and improved self- regulatory behaviors scores when evaluated at completion of the intervention and 6 and 12 months post intervention.

Aim 3 (Mediators): To test whether baseline traits and behaviors mediate the effect of AppCoach compared to App and Clinic.

Hypothesis 3: Higher baseline YFAS-c scores lower executive function scores and previous history with mobile platforms will mediate the efficacy of AppCoach and App.

Aim 4: To conduct a real-life economic analysis (costs, cost-savings and non-monetary benefits) of delivering AppCoach compared to 1) App and 2) Clinic.

Hypothesis 4: An addiction-based weight loss mHealth intervention will be more cost-effective than weight-loss coaching alone and in-person delivery of multidisciplinary weight-loss intervention.

Research Design Methods:

Study Design:

Multi-center, randomized, controlled, trial of an addiction based mobile health (mHealth) weight loss intervention plus personalized coaching (AppCoach) compared to receive 1)interactive addiction model based mHealth weight-loss intervention alone (App) and 2) Multidisciplinary in-clinic weight management program (Clinic).

Recruitment and Eligibility:

Study procedures will be approved by the Children's Hospital Los Angeles (CHLA), the Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center, Alta Med, UCLA, and Cedars Sinai Institutional Review Boards. Participants will be recruited for the intervention arms from newly referred patients of 5 interdisciplinary weight management clinics (CHLA, Alta Med, Los Angeles Biomedical Research Institute at Harbor-UCLA (LA Biomed), UCLA, and Cedars Sinai).

Patient Subjects:

Inclusion criteria include:

1. Age 14-18 years 2. Body mass index [BMI] ≥85th percentile for age and gender

Exclusion criteria include:

1. Concurrent participation in an alternative weight loss intervention
2. Blood pressure > 99th percentile for age, gender, and height
3. Known psychiatric illness and/or developmental delay
4. Participants Inability to read English

Parent Criteria:

1. Have an eligible child who meets the eligibility requirements listed above
2. Minimum age of 18 years old

Pre-Screening:

Clinic Recruitment:

Newly referred patients to the interdisciplinary clinics will be pre-screened for eligibility prior to their first clinic visit by an on-site clinical research coordinator (CRC). Those participants who meet eligibility criteria will be contacted via phone by the on-site CRC. The CRC will briefly introduce the study aims and intervention and request the youth and family to consider participation to be fully discussed at the first visit. The CRC will obtain the eligible participants' email address and send them a recruitment email.

Initial Visit:

1. On-site CRC will meet with eligible participants and provide details about the study procedures, obtain written consent from one parent/guardian and assent from each participant and answer any questions the participants and there parent may have.

   a. In order to standardize the study description, the CRC will first play an introductory video clip describing the study, the participant responsibilities and follow-up requirements.

   b. Upon obtaining verbal and written consent from one parent or guardian and verbal and written assent from each youth to participate in the study participants will be randomized to one of 3 intervention arms (AppCoach vs. App vs. Clinic)
2. All consenting participants will complete a battery of surveys (Refer to Measurements section).

   Covariates/Moderators:

   a. Yale Food Addiction Scale b. The Center for Epidemiologic Studies Depression scale c. The Perceived Stress Scale d. Behavior Rating Inventory of Executive function

   Outcomes:
   1. Intervention Satisfaction Survey
   2. The Adolescent Self-Regulatory Inventory (ASRI)
   3. Food Cravings Questionnaire
3. All consenting participants:

   1. AppCoach and App Groups will receive:

1. iPhones (as needed; participants will be required to have an iPhone). b. All Participants will receive: Wireless Bluetooth body weight scale (Wahoo Fitness Balance Scale; Wahoo fitness, Atlanta, GA) and a wireless Bluetooth digital food scale (Escali Smart Connect Kitchen Scale, Escali Corp., Burnsville, MN) both of which interfaced to the app.

c. Participants who require an iPhone will be loaned an iPhone 5S and accessories (including protective case), with an AT&T service plan for the duration of the study that includes: unlimited texting, unlimited plan, unlimited voice calls to and from other cell telephones, 700 voice call minutes for calls to and from landlines, unlimited night and weekend calls to and from landlines, International calls or texts including Canada are NOT allowed and not covered.

d. Participants will return the loaned phones at the completion of the intervention (Visit 3).

e. The referring provider will receive a letter informing them that the youth they referred to the weight management clinic will be participating in this study for 6 months and then will be offered enrollment back into the initial referral program is desired.

4. AppCoach Participants:

1. Each participant will register via a computer and then login with the app.
2. Participants will weigh-in on a scale in a private area and enter weight data on their iPhones.
3. On-site CRC will go through each section of app and have participants enter data.
4. Follow Up: Participants will schedule weekly 15 minute phone meetings with a coach and return for clinic visits at 3,6,12 and 18 months. The first phone visit will be via HIPAA secure video conferencing between the coach and the participant.

   5. App Participants:

a. Each participant will register via a computer and then login with the app. b. Participants will weigh-in on a scale in a private area and enter weight data on their iPhones.

c. On-site CRC will go through each section of app and have participants enter data.

d. Follow Up: Participants will schedule clinic visits at 3,6,12 and 18 months. 6. Clinic Participants:

1. Each participant will attend a multi-disciplinary in-clinic intervention that consists of 6 sessions (100 minutes for the first visit and 80 minutes for follow up visits).
2. They will travel to the local site of recruitment and attend 6 sessions in which they will meet with a provider team.
3. Participants will weigh-in on a scale in a private area and receive a wireless body and food scale
4. Follow Up: Participants will return clinic visits monthly for 6 months and then at 12 and 18 months post consent for maintenance follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age 14-18 years
* Body mass index [BMI] ≥85th percentile for age and gender

Exclusion Criteria:

* Concurrent participation in an alternative weight loss intervention
* Blood pressure > 99th percentile for age, gender, and height
* Known poorly controlled psychiatric illness and/or developmental delay
* Participants Inability to read English

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 161 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alaina Vidmar, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital of Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pretlow RA, Stock CM, Allison S, Roeger L. Treatment of child/adolescent obesity using the addiction model: a smartphone app pilot study. Child Obes. 2015 Jun;11(3):248-59. doi: 10.1089/chi.2014.0124. Epub 2015 Mar 11. PMID 25760813
- [Background] Tompkins CL, Laurent J, Brock DW. Food Addiction: A Barrier for Effective Weight Management for Obese Adolescents. Child Obes. 2017 Dec;13(6):462-469. doi: 10.1089/chi.2017.0003. Epub 2017 Jul 20. PMID 28727935
- [Background] Majeed-Ariss R, Baildam E, Campbell M, Chieng A, Fallon D, Hall A, McDonagh JE, Stones SR, Thomson W, Swallow V. Apps and Adolescents: A Systematic Review of Adolescents' Use of Mobile Phone and Tablet Apps That Support Personal Management of Their Chronic or Long-Term Physical Conditions. J Med Internet Res. 2015 Dec 23;17(12):e287. doi: 10.2196/jmir.5043. PMID 26701961
- [Background] Schulte EM, Gearhardt AN. Development of the Modified Yale Food Addiction Scale Version 2.0. Eur Eat Disord Rev. 2017 Jul;25(4):302-308. doi: 10.1002/erv.2515. Epub 2017 Mar 29. PMID 28370722
- [Derived] Metzendorf MI, Wieland LS, Richter B. Mobile health (m-health) smartphone interventions for adolescents and adults with overweight or obesity. Cochrane Database Syst Rev. 2024 Feb 20;2(2):CD013591. doi: 10.1002/14651858.CD013591.pub2. PMID 38375882
- [Derived] Pretlow R, Glasner S. Reconceptualization of eating addiction and obesity as displacement behavior and a possible treatment. Eat Weight Disord. 2022 Oct;27(7):2897-2903. doi: 10.1007/s40519-022-01427-1. Epub 2022 Jun 22. PMID 35731464
- [Derived] Vidmar AP, Yamashita N, Fox DS, Hegedus E, Wee CP, Salvy SJ. Can a Behavioral Weight-Loss Intervention Change Adolescents' Food Addiction Severity? Child Obes. 2022 Apr;18(3):206-212. doi: 10.1089/chi.2021.0271. Epub 2022 Jan 7. PMID 35006001
- [Derived] Lopez KE, Salvy SJ, Fink C, Werner J, Wee CP, Hegedus E, Gonzalez J, Fox DS, Vidmar AP. Executive Functioning, Depressive Symptoms, and Intervention Engagement in a Sample of Adolescents Enrolled in a Weight Management Program. Child Obes. 2021 Jun;17(4):281-290. doi: 10.1089/chi.2020.0334. Epub 2021 Apr 7. PMID 33826861
- [Derived] Vidmar AP, Salvy SJ, Pretlow R, Mittelman SD, Wee CP, Fink C, Steven Fox D, Raymond JK. An addiction-based mobile health weight loss intervention: protocol of a randomized controlled trial. Contemp Clin Trials. 2019 Mar;78:11-19. doi: 10.1016/j.cct.2019.01.008. Epub 2019 Jan 14. PMID 30654026

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Parents were not enrolled. Only adolescents provided informed consent to enroll in the study.
Groups:
- App Plus Coaching (AC): 6 month addiction model based weight loss intervention in the form of an iPhone app coupled with personalized coaching.
  App: a. 6 month app intervention: Problem Food Withdrawal, Snacking Elimination and Food Amount Reduction b. Daily Weigh In c. App based reminders d. Follow Up: Face-to-face clinic visits at 3,6,12 and 18 months.
  Coaching: a. 6 month addiction based intervention: Problem Food Withdrawal, Snacking Elimination and Food Amount Reduction.
  b. Daily Weighing c. Daily Text messages from Coach d. Weekly 15 minute phone meetings with Coach e. Follow Up: Face-to-face clinic visits at 3,6,12 and 18 months post consent
- App Alone (AA): 6 month addiction model based weight loss intervention in the form of an iPhone app.
  App: a. 6 month app intervention: Problem Food Withdrawal, Snacking Elimination and Food Amount Reduction b. Daily Weigh In c. App based reminders d. Follow Up: Face-to-face clinic visits at 3,6,12 and 18 months.
- Clinic: In-Clinic Multi-disciplinary monthly weight management program. Curriculum adapted from the KidsNFitness Program and administered by an MD, RD, Psychologist and Health Educator over 90 minute sessions
  Clinic: Modified KidsNFitness: a. 6 month in-clinic, evidence-based, multi-disciplinary intervention b. 90 minute sessions, in clinic that occur every month for 6 months c. Follow Up: Face-to-face clinic visits Monthly x 6 months followed by face-to-face visit at12 and 18 months.
Period: Overall Study
Arm/Group | App Plus Coaching (AC) | App Alone (AA) | Clinic
Started | 54 | 53 | 54
Completed | 37 | 23 | 42
Not Completed | 17 | 30 | 12

BASELINE CHARACTERISTICS:
Population: The baseline population is akin to those seen at CHLA and is as anticipated based on the cohort model that was accessed for recruitment.
Groups:
- Total: Total of all reporting groups
Arm/Group | App Plus Coaching (AC) | App Alone (AA) | Clinic | Total
Number analyzed (Participants) | 54 | 53 | 54 | 161
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 54 | 53 | 54 | 161
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 15 [14 to 17] | 16 [15 to 16] | 16 [14 to 17] | 16 [14 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 32 | 39 | 105
  Male | 20 | 21 | 15 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 29 | 28 | 77
  Not Hispanic or Latino | 34 | 24 | 26 | 84
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 54 | 53 | 54 | 161
Body Mass Index Z-score [Mean (Standard Deviation); unit: Z-score] — Body Mass Index (BMI) Z-score is derived from the World Health Organization (WHO) growth standards. A Z-score of 0 indicates the population mean BMI for a specific age and sex group based on the reference population. Z-scores greater than 0 indicate higher BMI values compared to the average of the reference population, which is associated with overweight or obesity. Z-scores less than 0 indicate lower BMI values, which may suggest underweight. Z-score ≥ 1: This indicates overweight status; Z-score ≥ 2: This indicates obesity; Z-score ≥ 3: This indicates severe obesity.
  Z-score | 2.2 (0.5) | 2.2 (0.5) | 2.3 (0.4) | 2.2 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: %BMIp95
Description: Mean change in excess BMI percent over the 95th percentile (%BMIp95) over the study period compared at 6 months to baseline. value at 6 months minus value at baseline
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | App Plus Coaching (AC) | App Alone (AA) | Clinic
Number analyzed (Participants) | 37 | 23 | 42
percent | -1.9 (1) | -1.2 (1.2) | -1.5 (2)

2. Secondary Outcome: Cost Analysis
Description: Real life economic analysis of the intervention arms compared to each other and in in-clinic intervention. The following data were collected throughout the study period to assess the implementation requirements (cost and labour) for each intervention arm: personnel time required for intervention implementation (including training time, visit time and preparation time), intervention specific equipment and maintenance, and cost of each activity per participant for the 6-month intervention period. A full cost-analysis evaluation of the intervention implementation is currently underway. Total accrued cost over the 6 month period compared to the other intervention.
Time Frame: 6 months
Population: Each groups' implementation cost was evaluated
Measure: Mean (Standard Deviation); unit: US dollars
Arm/Group | App Plus Coaching (AC) | App Alone (AA) | Clinic
Number analyzed (Participants) | 37 | 23 | 42
US dollars | 2076 (150) | 1122 (135) | 4034 (178)

3. Secondary Outcome: Yale Food Addiction Scale
Description: Yale Food Addiction Scale-Children (YFAS-c). The 25-tem scale assesses seven diagnostic criteria for substance dependence as it relates to eating. Items are answered on a 7-point Likert Scale ranging from 0 (never) to 7 (every day). Participants who report three or more symptoms and clinically significant impairment meet the criteria for food addiction (FA). The YFAS-c has shown good test-retest reliability. Reliability analyses have shown high internal consistency (Cronbach's alpha = 0.81) in the general paediatric population, and test-retest reliability between 0.79 and 0.84 in studies conducted in ethnically diverse paediatric populations.
  Total Score: The total score on the YFAS ranges from 0 to 11. A score of 0 indicates no symptoms of food addiction, while a score of 11 indicates the highest level of symptoms consistent with food addiction.
  Total Score Range: 0 to 11 Loss of Control Subscale Range: 0 to 5 Persistent Use Subscale Range: 0 to 6
Time Frame: 6 months
Population: YFAS-c was completed at baseline and throughout the study period. It has been well assessed in adolescents with obesity that up to 25-30% report positive YFAS-c scores consistent with addictive like eating behaviors.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | App Plus Coaching (AC) | App Alone (AA) | Clinic
Number analyzed (Participants) | 37 | 23 | 42
score on a scale | -0.5 [-0.5 to 0] | -0.5 [-1.5 to 0] | 0 [-1 to 0]

ADVERSE EVENTS:
Time Frame: 6 months
Description: Any unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research was assessed during the study period. Three types of adverse event data was collected: "All-Cause Mortality," "Serious," and "Other (Not Including Serious)" Adverse Events.
Arm/Group | App Plus Coaching (AC) | App Alone (AA) | Clinic
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/53 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/53 | 0/54
Other Adverse Events (participants affected / at risk) | 0/54 | 0/53 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-13): https://cdn.clinicaltrials.gov/large-docs/35/NCT03500835/Prot_SAP_000.pdf